CLINICAL TRIAL: NCT06505941
Title: Clinical Study on the Safety and Preliminary Efficacy of Umbilical Cord Mesenchymal Stem Cell Intravenous Infusion Therapy for Acute Respiratory Distress Syndrome
Brief Title: Clinical Study on the Safety and Preliminary Efficacy of hUC-MSCs Intravenous Infusion Therapy for ARDS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southeast University, China (Other)
Collaborators: Zhongda Hospital (Other); Yinguan Biologics, Shenzheng (Unknown)
Responsible Party: Principal Investigator, Jianfeng Xie, deputy director, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019ZDSYLL077-P06
Record Dates: First submitted 2024-04-02; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: acute respiratry distress syndrome; human umbilical cord derived mesenchymal stem cell; clinical study
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Carboxylesterase

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): 1 intravenous infusion of an equal volume of cell-free placebo.
  Interventions: Drug: Placebo
- MSC (Experimental): Name：Human umbilical cord mesenchymal stem cells Specification: 30 ml/bag Dosage: 1×106cells/kg, 5×106cells/kg, 10×106cells/kg Usage: Intravenous infusion The stem cells used in this study are human umbilical cord mesenchymal stem cells (hUC-MSCs), which are derived from umbilical cords donated by healthy mothers who have given birth in maternity hospitals. hUC-MSCs are extracted, processed, cultured and harvested from umbilical cord donors recruited by laboratories complying with the GMP standards. hUC-MSCs cell suspensions that have passed the quality control will be put into bags and transported to the hospitals for use by the subjects of the present clinical study.
  Interventions: Drug: umbilical cord mesenchymal stem cell

INTERVENTIONS:
Drug: umbilical cord mesenchymal stem cell — umbilical cord mesenchymal stem cell
  Other Names: cell
  Arms: MSC
Drug: Placebo — non-cell-containing placebo
  Arms: placebo

SUMMARY:
The object of this study is to observe the safety of umbilical cord mesenchymal stem cell therapy for acute respiratory distress syndrome, consisting with two phases.

DETAILED DESCRIPTION:
The secondary objectives are to observe the preliminary efficacy of umbilical cord mesenchymal stem cell therapy for acute respiratory distress syndrome. Phase One is an open-label, dose-escalation clinical study. Following safety and tolerability conclusions from Phase One, and upon evaluation and approval by the data safety committee and ethics committee, conduct Phase Two study, which will be a randomized, double-blind, placebo-controlled study. Dosage selection will be based on the safest and most effective dosage determined from Phase One results.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years, regardless of gender;
2. Meeting the ARDS Berlin diagnostic criteria;
3. Definite diagnosis within 72 hours;
4. P/F < 150mmHg;
5. Understanding and signing informed consent.

Exclusion Criteria:

1. Women of childbearing potential with a positive serum pregnancy test before medication, pregnant women, or lactating women;
2. ARDS directly caused by physical or chemical factors;
3. Moderate to severe liver damage (Child-Pugh score >12);
4. Chronic heart failure, New York Heart Association functional class IV;
5. Severe kidney disease undergoing renal replacement therapy;
6. Severe lung disease, Grade III or IV pulmonary hypertension, receiving oxygen therapy or ventilator support for more than one month in the six months prior to screening, end-stage lung disease, or severe physical limitations due to chest wall deformity;
7. Immunodeficiency, receiving immunosuppressive therapy within 2 weeks (except for low-dose corticosteroids), or with lymphoma, leukemia, or acquired immune deficiency syndrome; history of organ transplantation, bone marrow transplantation, or autologous hematopoietic stem cell suppression;
8. Expected survival time of less than 48 hours due to terminal illness;
9. Patients diagnosed with deep vein thrombosis (DVT) or pulmonary embolism (PE) in the past three months;
10. Patients receiving ECMO therapy;
11. Hepatitis B, hepatitis C, syphilis, or HIV infection.
12. eGFR < 30ml/min/BSA;
13. ALT > 5 × ULN;
14. Absolute neutrophil count < 1500/μL;
15. Subjects who have participated in other clinical studies within the past month (excluding those who have not received intervention), or are currently participating in other experimental treatments;
16. Subjects deemed unlikely to benefit from the study by the investigator, or deemed unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
The safety of umbilical cord mesenchymal stem cell therapy for acute respiratory distress syndrome. | The 1, 6, 24 hours; 3、7、14、21 days and 4, 12, 24, 36, 48 weeks after injection.
  The 28-day mortality of patients receiving umbilical cord mesenchymal stem cell therapy

SECONDARY OUTCOMES:
The efficacy of umbilical cord mesenchymal stem cell therapy for acute respiratory distress syndrome. | The 1, 6, 24 hours; 3、7、14、21 days and 4, 12, 24, 36, 48 weeks after injection.
  Oxygenation index situation change (PaO2/FiO2) of patients receiving umbilical cord mesenchymal stem cell therapy

IPD SHARING:
Plan to Share IPD: No